CLINICAL TRIAL: NCT05301868
Title: A Multicenter Clinical Study to Evaluate the Efficacy and Feasibility of a 24-week Multidomain Intervention Via a None-face-to-face Platform in Mild Cognitive Impairment
Brief Title: Multidomain Intervention Via a None-face-to-face Platform in Mild Cognitive Impairment
Acronym: EXTENDED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Seong Hye Choi, MD, Professor, Inha University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-02-009
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidomain intervention (Experimental): The participants in the intervention arm will receive all five components of the intervention: (1) monitoring and management of metabolic and vascular risk factors; (2) cognitive training; (3) physical exercise; (4) nutritional guidance; and (5) motivational training via none-face-to-face tablet PC application (app).
  Interventions: Behavioral: Multidomain intervention

INTERVENTIONS:
Behavioral: Multidomain intervention — For 24 weeks, participants will receive cognitive training twice a week, exercise 3 times a week, nutrition education 12 times, and education about vascular risk factor management every 2 weeks using the tablet PC application.
  Other Names: multidomain cognitive intervention

SUMMARY:
This study will be done to investigate the feasibility and effectiveness of a 24-week multidomain intervention program consisting of cognitive training, exercise, nutrition management, vascular disease risk factor management, and motivational enhancement on the cognitive function via none-face-to-face platform in mild cognitive impairment.

DETAILED DESCRIPTION:
The physical exercise program will consist of aerobic exercise, exercise to enhance balance and flexibility, muscle-strengthening activities involving major muscle groups, and finger-toe movements. Cognitive training targets the cognitive domains of episodic memory, executive function, attention, working memory, calculation, and visuospatial function. Cognitive training will be conducted using a tablet-based application. Participants will be advised to eat something according to the recommendation of the Mediterranean-DASH Intervention for Neurodegenerative Delay diet (MIND) diet. They will be educated about vascular risk factor management every 2 weeks. The purpose of the motivational enhancement program is to induce, maintain, and strengthen motivation, which is a psychological resource to help maintain dementia prevention activities. All intervention will be administered via tablet personal computer (PC) application at home.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed end-of-study evaluation and participated in the preceding randomized controlled trial (RCT) "Multidomain Interventions Via Face-to-face and Video Communication Platforms in Mild Cognitive Impairment".
* Being able to use the tablet PC through education, or having a person who can help a participant use the tablet PC.
* Having a reliable informant who could provide investigators with the requested information
* Provide written informed consent

Exclusion Criteria:

* Major psychiatric illness such as major depressive disorders
* Dementia
* Other neurodegenerative disease (e.g., Parkinson's disease)
* Malignancy within 5 years
* Cardiac stent or revascularization within 1 year
* Serious or unstable symptomatic cardiovascular disease
* Other serious or unstable medical disease such as acute or severe asthma, active gastric ulcer, severe liver disease, or severe renal disease
* Severe loss of vision, hearing, or communicative disability
* Any conditions preventing cooperation as judged by the study physician
* Significant laboratory abnormality that may result in cognitive impairment
* Illiteracy
* Unable to participate in exercise program safely
* Coincident participation in any other intervention trial

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of cognition | Change from Baseline at 24 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status

SECONDARY OUTCOMES:
Change of global cognition | Change from Baseline at 24 weeks
  Mini-Mental State Examination (range 0-30). Higher scores indicate better performance.
Change of function | Change from Baseline at 24 weeks
  Clinical Dementia Rating scale-Sum of Boxes (range 0-18). Higher scores indicate worse performance.
Change of subjective memory | Change from Baseline at 24 weeks
  Prospective and Retrospective Memory Questionnaire (range 16-80). Higher scores indicate worse performance.
Change of depression | Change from Baseline at 24 weeks
  Geriatric Depression Scale-15 items (range 0-15). Higher scores indicate worse performance.
Quality of life assessed by the Quality of life-Alzheimer's disease | Change from Baseline at 24 weeks
  Quality of life-Alzheimer's disease (range 0-52). Higher scores indicate better performance.
Change of activities of daily living | Change from Baseline at 24 weeks
  Bayer Activities of Daily Living (range 1-10). Higher scores indicate worse performance.
Change of nutritional behavior | Change from Baseline at 24 weeks
  Nutrition Quotient for elderly (range 0-100). Higher scores indicate better performance.
Change of nutrition | Change from Baseline at 24 weeks
  Mini Nutritional Assessment (range 0-14). Higher scores indicate better performance.
Change of motor function | Change from Baseline at 24 weeks
  Short Physical Performance Battery (range 0-12). Higher scores indicate better performance.
Sleep quality assessed by the Pittsburgh Sleep Quality Index | Change from Baseline at 24 weeks
  Pittsburgh Sleep Quality Index (range 0-21). Higher scores indicate worse performance.
Change of motivation | Change from Baseline at 24 weeks. Higher scores indicate better performance.
  Self Determination Index (SDI) (range -66~66). Higher scores of SDI indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hye Choi, MD, PhD, Principal Investigator — Inha University Hospital
Locations (4):
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Ewha Womans Seoul Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 2 years since March 2024.
Access Criteria: Reasonable request